CLINICAL TRIAL: NCT04446923
Title: Surgical Hand Antisepsis With Propan-ol-1 60% Per Rubbing and Scrubbing in Accordance With European Norm Regulation 12791
Brief Title: Surgical Hand Antisepsis With Propan-ol-1 60% Per Rubbing and Scrubbing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RICBEC1-UCM
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Skin Diseases; Surgical Site Infection
Keywords: hand antisepsis
MeSH Terms: conditions — Skin Diseases; Surgical Wound Infection | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Crossover design is used
Who Masked: Outcomes Assessor
Masking Description: The samples will be sent to the laboratory with numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand antisepsis by scrub (Experimental): Hand antisepsis by scrub using propan-ol-1 60%
  Interventions: Drug: Hand antisepsis by scrub
- Hand antisepsis by rub (Active Comparator): Hand antisepsis by rub using propan-ol-1 60%
  Interventions: Drug: Hand antisepsis by scrub

INTERVENTIONS:
Drug: Hand antisepsis by scrub — Surgical Hand scrubbing using P-1 of both hands using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side.
  Other Names: Propanolol
  Arms: Hand antisepsis by scrub
Drug: Hand antisepsis by scrub — Surgical Hand rubbing using P-1 of both hands using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side.
  Other Names: Propanolol
  Arms: Hand antisepsis by rub

SUMMARY:
The present study evaluates the effects of to compare bactericidal efficacy using the reference antiseptic product propan-ol-1 60% using the hand rub method versus hand scrub method in order to test if pass the standard european norm 12791.

DETAILED DESCRIPTION:
The investigators conducted a crossover clinical trial to evaluate the antiseptic effectiveness of preoperative surgical scrubbing using propan-ol-1 60% by rub and scrub. Samples will be taken from the hands of each volunteer after a surgical hands antiseptic.

ELIGIBILITY:
Inclusion Criteria:

* Participants without systemic pathologies, with healthy skin of the hands and short fingernails.
* They do not use substances with antibacterial action.

Exclusion Criteria:

* Taken antibiotics before 10 days of the intervention.
* Wear any jewellery on the hands.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Reduction of bacterial load immediately after hand scrub | Change from bacterial load at 5 minutes.
  Participants will scrub the liquid vigorously from hand to the wrists according with the standard handrub procedure.

SECONDARY OUTCOMES:
Reduction of bacterial load after 3 hours of hand scrub | Change from bacterial load at 3 hours.
  Participants will scrub the liquid vigorously from hand to the wrists according with the standard handrub procedure after 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Becerro de Bengoa Vallejo, PhD, Principal Investigator — Ricardo becerro de Bengoa Vallejo
Locations (1):
- Ricardo Becerro de Bengoa Vallejo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
A number will be assigned to each participant